CLINICAL TRIAL: NCT06143501
Title: Alterations in Intestinal Microbiota, Metabolites, and Immune Cells Pre- and Post-Transplantation of Allogeneic Hematopoietic Stem Cells
Brief Title: Alterations in Intestinal Microbiota, Metabolites, and Immune Cells in Allo-HSCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Other Study IDs: Pre-Post Allo-HSCT Monitoring
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Graft Vs Host Disease
Keywords: Allo-HSCT; Intestinal Microbiota; Metabolites; Immunity
MeSH Terms: conditions — Graft vs Host Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Allo-HSCT Recipients
  Interventions: Diagnostic Test: Blood Sample; Diagnostic Test: Stool Sample; Diagnostic Test: Urine Sample
- Healthy Volunteers
  Interventions: Diagnostic Test: Blood Sample; Diagnostic Test: Stool Sample; Diagnostic Test: Urine Sample

INTERVENTIONS:
Diagnostic Test: Blood Sample — 6 ml blood (collection occurs once pre-transplantation and at three designated follow-up time points post-transplantation)
Diagnostic Test: Stool Sample — pea-sized amount (collection occurs once pre-transplantation and at three designated follow-up time points post-transplantation)
Diagnostic Test: Urine Sample — 8 ml (collection occurs once pre-transplantation and at three designated follow-up time points post-transplantation)

SUMMARY:
This research project delves into the critical role of gut immunity in the occurrence and progression of acute graft-versus-host disease (aGVHD) post allogeneic hematopoietic stem cell transplantation (allo-HSCT). Addressing the current gaps in understanding the involvement of intestinal microbiota, metabolites, and cellular metabolism in clinical aGVHD, the study involves comprehensive analyses on 200 allo-HSCT patients and 50 healthy volunteers. By scrutinizing changes in gut microbiota, metabolites, and immune cell metabolism, the research aims to shed light on their roles in allo-HSCT and their correlation with post-transplant complications. The findings are poised to offer crucial insights for diagnosing and prognosticating complications following transplantation.

DETAILED DESCRIPTION:
The intestinal immune system plays a pivotal role in the onset, progression, and evolution of acute graft-versus-host disease (aGVHD) following allogeneic hematopoietic stem cell transplantation (allo-HSCT). However, the precise contributions and mechanisms underlying the involvement of intestinal microbiota, metabolites, and cellular metabolism in immune regulation during clinical aGVHD remain unclear.

This research initiative aims to collect peripheral blood, fecal, and urine samples from 200 patients before and after transplantation as well as 50 healthy volunteers. Comprehensive analyses, including metagenomics, 16S rRNA sequencing, transcriptomics, metabolomics, single-cell sequencing, as well as assessments of immune cell function and inflammatory cytokines, will be conducted. Additionally, longitudinal follow-up observations will be performed to monitor post-transplant complications, relapse and immune reconstitution.

By investigating the dynamics of gut microbiota, metabolites, and cellular metabolism and analyzing their correlation with changes in immune responses, this study seeks to elucidate the roles of intestinal microbiota, metabolites, and immune cell metabolism in the context of allo-HSCT. The findings are anticipated to provide insights into the correlation between these factors and outcomes of allo-HSCT patients, contributing valuable evidence for the diagnosis and prognosis assessment of complications following transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematologic disorders undergoing allo-HSCT.

Exclusion Criteria:

* Patients with confirmed pathogenic intestinal infections and severe systemic infections at the time of sampling.
* Diagnosis of autoimmune diseases, metabolic disorders, and chronic gastrointestinal diseases.
* Pre-transplant diseases not in complete remission.
* Post-transplant hematopoietic engraftment failure or pre-engraftment mortality.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Hematological patients will receive allo-HSCT in short time.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Complications | 2 years
  Recording and monitoring the occurrence of complications such as infection, GVHD, etc., documenting their onset time, type, severity, and management.
Relapse | 2 years
  Documenting and monitoring the occurrence of relapse in study subjects, including recording the time of onset, severity, and management.
Overall Survival | 2 years
  OS will be assessed from the first day of stem cells infused to death or last follow-up.

SECONDARY OUTCOMES:
Immune Function | Measured 3 months after stem cells infused
  Incidence of neutrophil recovery; Incidence of lymphocyte and monocyte subset recovery

CONTACTS AND LOCATIONS:
Overall Officials: Yang Xu, M.D, Study Chair — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No